CLINICAL TRIAL: NCT07207759
Title: MILLENIA: MultIpLe Long-tErm Conditions in Pregnancy aNd Experiences of mIdwifery cAre
Brief Title: MultIple Long-term Conditions in Pregnancy and Experiences of Midwifery Care
Acronym: MILLENIA
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Lancashire Teaching Hospitals NHS Foundation Trust (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 323932
Record Dates: First submitted 2025-06-12; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: How Pregnant and Postnatal Women With Two or More Long-term Health Conditions Experience Midwifery Care as Part of Multi-disciplinary Maternity Care
Keywords: Multiple Long-term Conditions; Midwife; Midwifery; Models of care; Multi-disciplinary care; Continuity of care(r); Healthcare use; Care experiences; Burden of treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interview participants: Up to 20 women or birthing people who are pregnant or have experienced pregnancy with two or more long-term health conditions in the last two years.
  Up to 20 midwives who provide care or manage services for women with two or more long-term health conditions or healthcare professionals who collaborate with midwives
- Co-design workshop participants: Up to 40 co-design participants including women and birthing people with two or more long-term health conditions who are pregnant or postnatal or have given birth in the last 3 years; partners/supporters/significant others of women with two or more long-term health conditions who are pregnant or postnatal or have given birth in the last 3 years; National Health Service maternity staff including midwives and healthcare professionals who provide care or manage services for women with two or more long-term health conditions; members of the Patient and Public Involvement and Engagement Group and Project Advisory Group; representatives from the study third sector Patient and Public Involvement and Engagement partners (Maternal Mental Health Alliance, Action on Pre-eclampsia and Social Action for Health); representatives from other relevant third sector organisations; health policy makers and commissioners

SUMMARY:
This is a qualitative study using in-depth semi-structured interviews. This study will explore pregnant women with two or more long-term health condition's (MLTC) experience of midwifery care and midwives and health professionals experience of providing midwifery care and multidisciplinary maternity care. This will be considered in relation to Treatment Burden and Minimally Disruptive Healthcare theories. This will be followed by co-design of guidance for midwifery care of pregnant women with MLTC. The aim is to develop a rich understanding of the topic and participant's lived experiences, to enable development of a resource which is meaningful to the key stakeholders. The study is part of a wider mixed methods study.

ELIGIBILITY:
Inclusion Criteria:

Interviews

Women and birthing people

* Women and birthing people with two or more pre-existing long-term health conditions (see appendix one) who are pregnant or postnatal or have given birth in the last 2 years
* Able to provide consent
* Able to participate in English or through an interpreter
* Age 18 or over Midwives and maternity health care professionals NHS maternity staff including midwives and healthcare professionals who provide or manage care for women with two or more long-term health conditions e.g., obstetricians, obstetric physicians, medicine, perinatal mental health, and primary care.

Co-design meetings

* Women and birthing people with two or more long-term health conditions who are pregnant or postnatal or have given birth in the last 3 years (to include those who have given birth in the last 2 years at the beginning of the study who participated in an interview
* Partners/supporters/significant others of women with two or more long-term health conditions who are pregnant or postnatal or have given birth in the last 3 years
* Able to provide consent
* Able to participate in English or through an interpreter
* Age 18 or over
* NHS maternity staff including midwives and healthcare professionals who provide care or manage services for women with two or more long-term health conditions
* Members of the Patient and Public Involvement and Engagement Group and Project Advisory Group
* Representatives from the study third sector partners (Maternal Mental Health Alliance, Action on Pre-eclampsia and Social Action for Health)
* Representatives from other relevant third sector organisations
* Health policy makers and commissioners

Exclusion Criteria:

Interviews Women and birthing people

* Women and birthing people without two or more pre-existing long-term health conditions
* Those who are not pregnant or have not given birth in the last two years
* Those who refuse or are unable to give consent
* Age under 18
* Age over 60

Midwives and maternity health care professionals NHS maternity staff including midwives and healthcare professionals who do not provide or manage care for women with two or more pre-existing long-term health conditions Co-design meetings

* Those who refuse or are unable to give consent
* Age under 18

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interviews: Women and staff with a range of physical and mental health long term conditions. Midwives and maternity healthcare professionals who provide care for women with MLTC such as obstetricians, obstetric physicians, or those in medicine, perinatal mental health and primary care.
  Co-design meetings: Some participants will be purposefully sampled from those who participated in interviews. If the desired sample size is not met through those participating in interviews, a further purposive sample will be recruited through third sector and professional networks and direct approach of potential participants at each site.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Experiences of care | 2025-2027
  Pregnant and postnatal women with two or more long-term health conditions experience of midwifery care, as part of multi-disciplinary maternity care

SECONDARY OUTCOMES:
Experiences of providing care | 2025-2027
  Midwives' experience of providing care for pregnant, birthing, and postnatal women with MLTC
Experiences of providing care | 2025-2027
  Health professionals experience of providing care for pregnant, birthing, and postnatal women with MLTC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://arc-sl.nihr.ac.uk/research-and-implementation/our-research-areas/maternity-and-perinatal-mental-health/exploring-0